CLINICAL TRIAL: NCT04036825
Title: Effectivity of Liquid Nutritional Supplementation in Improving Nutritional Status of Hospitalized Malnutrition Patients: A Single-Blind Randomized Controlled Trial
Brief Title: Liquid Nutritional Supplement on Malnutrition Hospitalized Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Marcellus Simadibrata, Prof. PhD., SpPD, KGEH, Prof. dr. Marcellus Simadibrata, Ph.D., SpPD-KGEH, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-01-0082
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Malnutrition
Keywords: Liquid Nutritional Supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid Nutritional Supplement from Hospital Product (Experimental): This group received liquid nutritional supplement from hospital product. The product is in a form of low lactose milk ready to drink with volume 200 ml and will be given 2 times daily for 14 days. This product is consist of 1.017 kcal/ml, 10 vitamin and 9 mineral
  Interventions: Dietary Supplement: Liquid Nutritional Supplement from Hospital Product
- Placebo (Placebo Comparator): This group received standard liquid nutritional supplement as a placebo. Placebo will be given 2 times daily for 14 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Liquid Nutritional Supplement from Hospital Product — Liquid Nutritional Supplement from Hospital Product is given 2 times daily for 14 days
  Arms: Liquid Nutritional Supplement from Hospital Product
Dietary Supplement: Placebo — Standard nutritional supplement is given 2 times daily as placebo for 14 days
  Arms: Placebo

SUMMARY:
The aim of this study is to know the effectivity of liquid nutritional supplementation in malnutrition hospitalized patients

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years old to 60 years old
* malnutrition hospitalized patient based on European Society for Clinical Nutrition and Metabolism (ESPEN) 2015 criteria
* agreed to participate

Exclusion Criteria:

* malignancy
* chronic kidney disease stage III-V
* decompensated hepatic cirrhosis
* allergic to milk or lactose intolerance
* could not be randomised and participate in this study by clinical judgement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of Body Mass Index (BMI) | 0 and 14 days
  BMI was assessed from height and body calculation. Classification of BMI is based on World Health Organization (WHO) classification.

SECONDARY OUTCOMES:
Change of Subjective Global Assessment (SGA) rank | 0 and 14 days
  SGA rank is classified to A (well nourished), B (moderately malnourished) and C (severely malnourished) and these option are chosen based on history and physical examination that are stated in the SGA form.
Change of body fat percentage | 0 and 14 days
  Body fat percentage is assessed by Bioelectrical Impedance Analysis (BIA)
Change of handgrip strength test score | 0 and 14 days
  Handgrip strength is assessed by handgrip strength score.
Change of hemoglobin level | 0 and 14 days
  Hemoglobin level is obtain from laboratory test
Change of prealbumin level | 0 and 14 days
  Prealbumin level is obtain from laboratory test
Change of Blood Urea Nitrogen (BUN) level | 0 and 14 days
  BUN level is obtain from laboratory test
Change of lipid profile level | 0 and 14 days
  Lipid profile level is obtain from laboratory test
Change of blood glucose level | 0 and 14 days
  Blood glucose level is obtain from laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Marcellus Simadibrata, Principal Investigator — Division Of Gastroenterology Department Of Internal Medicine Faculty Of Medicine Universitas Indonesia
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta Pusat, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT04036825/Prot_SAP_001.pdf